CLINICAL TRIAL: NCT01612884
Title: Antiplatelet Therapy Guided by Thrombelastography in Patients With Acute Coronary Syndromes (TEGCOR Study)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Rolf Kreutz, M.D., Associate Professor of Clinical Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1106005745
Record Dates: First submitted 2012-06-04; First posted 2012-06-06 (Estimated); Results first posted 2018-04-26 (Actual); Last update posted 2018-04-26 (Actual); Status verified 2018-03

CONDITIONS: Thrombosis; Coronary Artery Disease
MeSH Terms: conditions — Thrombosis; Coronary Artery Disease | interventions — Prasugrel Hydrochloride; Clopidogrel

ARMS (2):
- TEG (Other): Clopidogrel non-response defined as MA≥69 Clopidogrel response defined as MA<69
  Interventions: Drug: Prasugrel; Drug: Clopidogrel
- Light transmittance aggregometry (Other): Clopidogrel non-response defined as MPA ADP >42.9% Clopidogrel response defined as MPA ADP <42.9%
  Interventions: Drug: Prasugrel; Drug: Clopidogrel

INTERVENTIONS:
Drug: Prasugrel — Prasugrel 60mg loading dose at time of PCI if clopidogrel non-responder
Drug: Clopidogrel — Clopidogrel 300mg loading dose at time of PCI if clopidogrel responder

SUMMARY:
Personalized treatment approaches and antiplatelet drug choice have been proposed to optimize safety of coronary stenting by reducing heart attacks and repeat interventions while simultaneously minimizing adverse bleeding events. This study compares the efficacy of two laboratory guided treatment algorithms to personalize antiplatelet medication choice after coronary stenting

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted with acute coronary syndrome (unstable angina, non-ST elevation myocardial infarction) and referred for coronary angiography.
* Current therapy with clopidogrel (at least 300mg loading dose, or 75mg po daily for >5 days)
* Age range 21-75 years.

Exclusion Criteria:

* Unable to give consent
* Age younger than 21 years, greater than 75 years
* History of stroke
* Body weight <60 kg
* Acute STEMI,
* Thrombocytopenia<100'000,
* requirement for chronic warfarin therapy

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2011-08; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Eskenazi Health, Indianapolis, Indiana
  - Indiana University Health Methodist Hospital, Indianapolis, Indiana

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 67 subjects were enrolled and underwent testing on day 0. Only 37 of those subjects underwent PCI, and therefore were randomized to either LTA or TEG guided intervention arm. The remainder of subjects were treated medically without PCI or were referred for CABG (see flow diagram in protocol) and did not get randomized to any intervention arm.
Groups:
- Thrombelastography (TEG) Guided: Clopidogrel non-response defined as MA≥69 Clopidogrel response defined as MA<69
  Prasugrel: Prasugrel 60mg loading dose at time of PCI if clopidogrel non-responder
  Clopidogrel: Clopidogrel 300mg loading dose at time of PCI if clopidogrel responder
- Light Transmittance Aggregometry Guided: Clopidogrel non-response defined as MPA ADP >42.9% Clopidogrel response defined as MPA ADP <42.9%
  Prasugrel: Prasugrel 60mg loading dose at time of PCI if clopidogrel non-responder
  Clopidogrel: Clopidogrel 300mg loading dose at time of PCI if clopidogrel responder
Period: Overall Study
Arm/Group | Thrombelastography (TEG) Guided | Light Transmittance Aggregometry Guided
Started | 19 | 18
Completed | 19 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Thrombelastography (TEG) Guided | Light Transmittance Aggregometry Guided | Total
Number analyzed (Participants) | 19 | 18 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (9.8) | 53.2 (10.5) | 54.2 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 10 | 15
  Male | 14 | 8 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 8 | 22
  White | 5 | 10 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 18 | 37

OUTCOME MEASURES:

1. Primary Outcome: Thrombelastography (TEG) MA
Description: Persistence of high tensile clot strength measured by TEG 16-24 hours after reloading of either clopidogrel or prasugrel
Time Frame: 1 day
Population: TEG-MA (mm) at 16-24 hours outcome measure
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Thrombelastography (TEG) Guided | Light Transmittance Aggregometry Guided
Number analyzed (Participants) | 19 | 18
mm | 66.4 (11) | 65.8 (6.9)
Statistical Analysis 1: Comparison: Thrombelastography (TEG) Guided vs Light Transmittance Aggregometry Guided; Test type: Other — Student's T-test; p = 0.85, t-test, 2 sided

2. Secondary Outcome: Number of Participants With Ischemic Events
Description: Death, recurrent myocardial infarction, recurrent unstable angina, repeat coronary intervention
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Thrombelastography (TEG) Guided | Light Transmittance Aggregometry Guided
Number analyzed (Participants) | 19 | 18
Participants
  Death: Event | 0 | 0
  Death: No Event | 19 | 18
  Myocardial Infarction: Event | 1 | 0
  Myocardial Infarction: No Event | 18 | 18
  Recurrent coronary intervention: Event | 3 | 2
  Recurrent coronary intervention: No Event | 16 | 16
  Unstable Angina: Event | 2 | 2
  Unstable Angina: No Event | 17 | 16
Statistical Analysis 1: Comparison: Thrombelastography (TEG) Guided vs Light Transmittance Aggregometry Guided; Test type: Other — Chi-Square; p = 0.93, Chi-squared

3. Secondary Outcome: Number of Participants With Bleeding Events
Description: Major or Minor Bleeding according to TIMI criteria
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Thrombelastography (TEG) Guided | Light Transmittance Aggregometry Guided
Number analyzed (Participants) | 19 | 18
Participants
  Bleeding | 0 | 0
  No Bleeding | 19 | 18
Statistical Analysis 1: Comparison: Thrombelastography (TEG) Guided vs Light Transmittance Aggregometry Guided; Test type: Other — Chi-Square; p > 0.05, Chi-squared

ADVERSE EVENTS:
Time Frame: Complete duration of study period (6 months)
Arm/Group | Thrombelastography (TEG) Guided | Light Transmittance Aggregometry Guided
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 0/19 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2011-04-11): https://cdn.clinicaltrials.gov/large-docs/84/NCT01612884/Prot_000.pdf
  • Statistical Analysis Plan (2011-04-11): https://cdn.clinicaltrials.gov/large-docs/84/NCT01612884/SAP_001.pdf